CLINICAL TRIAL: NCT00797693
Title: Oral Versus Vaginal Misoprostol as Cervical Ripening Agent Prior to Surgical Termination of First Trimester Missed Abortions in Hawler Maternity Teaching Hospital in Erbil/Iraq
Brief Title: Misoprostol in Termination of First Trimester Missed Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Collaborators: HAWLER Maternity Hospital (Unknown)
Responsible Party: Scientific Committe, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 324/2
Record Dates: First submitted 2008-11-21; First posted 2008-11-25 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: Miscarriage
Keywords: First trimester; missed abortion; misoprostol; cervical ripening; oral; vaginal; first trimester missed abortion
MeSH Terms: conditions — Abortion, Spontaneous; Abortion, Missed | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaginal Misoprostol (Experimental): A drug is given vaginally and to compare this with an oral administration of the same drug to find it is effect on it is effect on the cervix
  Interventions: Drug: Misoprostol ( Cytotec) 200 microgram a tablet
- Oral Misoprostol (Experimental): A drug is given vaginally and to compare this with an oral administration of the same drug to find it is effect on it is effect on the cervix
  Interventions: Drug: Misoprostol ( Cytotec) 200 microgram a tablet

INTERVENTIONS:
Drug: Misoprostol ( Cytotec) 200 microgram a tablet — In this study, two arms we put under study ... and to find how far a single drug, Misoprostol, is effective to have changes on the cervix.
  Other Names: PHARMACIA CORPORATION - Istanbul, serial number 022-00; 200 microgram a tablet

SUMMARY:
The purpose of this study is to determine whether oral versus vaginal misoprostol is effective in termination of first trimester missed abortion and to compare between two different routes.

DETAILED DESCRIPTION:
Objective: To compare the effectiveness of oral versus vaginal misoprostol prior to surgical termination of first trimester missed abortion as cervical priming agent , the difference of cervical dilatation immediately prior to operation , the duration of operation and side effects between two treatment groups.

Design: This study was conducted as randomised study.

Setting: Maternity Teaching Hospital in Hawler/ Kurdistan/ Iraq.

Population: Over a period of six months from the first of January to the thirtieth of June, 2008, one hundred women were included in this study. They were cases of first trimester abortion (6-12 weeks).

Method: Patients were randomly selected for the type of treatment they received. The first group (oral) were assigned to receive 400 micrograms of misoprostol orally as preoperative cervical priming agent, where as the second group (vaginal) were allocated to have treatment either with vaginal misoprostol to receive 400 micrograms vaginally.

Main outcome measure: Oral versus vaginal misoprostol as cervical ripening agent prior to termination of first trimester missed abortion.

Keywords: First trimester, missed abortion, misoprostol, cervical ripening, oral, vaginal.

ELIGIBILITY:
Inclusion Criteria:

* All patients were cases of first trimester missed abortion.
* They have uneventful history apart from history of slight vaginal bleeding, with normal general examination. Gynecological examination revealed no vaginal bleeding or discharge with no dilatation of the internal os with enlarged uterus.

Exclusion Criteria:

* Cases with suspected or proven ectopic pregnancy, history of Caesarean section, medical diseases, a known hypersensitivity to a drug, smokers, patients with abnormal results of investigation and the presence of vaginal bleeding were excluded from the study.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Priming with misoprostol administered orally or vaginally three hours before surgical termination of first trimester missed abortion under general anesthesia facilitates cervical dilatation | 6 months

SECONDARY OUTCOMES:
Higher patient satisfaction for self administered oral misoprostol at home | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Maternity Teaching Hospital, Erbil, Hawler, Iraq